CLINICAL TRIAL: NCT00757705
Title: An Open-label Prospective Trial to Evaluate the Tolerability, Safety and Maintained Efficacy of a Transition to Paliperidone ER in Subjects With Schizophrenia Previously Unsuccessfully Treated With Other Oral Antipsychotics
Brief Title: An Efficacy, Safety And Tolerability Study of Flexibly Dosed Paliperidone Extended-Release (ER) in Participants With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014308; R076477SCH4033
Record Dates: First submitted 2008-09-19; First posted 2008-09-23 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone Extended-Release
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone Extended-Release (ER) (Experimental)
  Interventions: Drug: Paliperidone ER

INTERVENTIONS:
Drug: Paliperidone ER — Participants will receive paliperidone ER tablet in dose range of 3 to12 milligram (mg) per day orally once daily for 24 weeks as per Investigator's discretion based on the individual participant's clinical response to and tolerability of the study drug.
  Other Names: R076477; Invega

SUMMARY:
The purpose of the study is to explore the maintained efficacy, tolerability, and safety of flexibly dosed paliperidone extended-release (ER) in participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self) previously unsuccessfully treated with other oral atypical antipsychotic medication.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), non-randomized (the study drug is not assigned by chance), single arm, multicenter (when more than one hospital or medical school team work on a medical research study), 24-week study. Participants can be transitioned to an effective dose of paliperidone ER from any oral antipsychotic medication without the need for titration due to lack of efficacy, lack of tolerability or safety, lack of compliance or other reason. A transition period of maximum 4 weeks will be allowed. Throughout the study, participants will receive flexible dose of 3 to 12 milligram (mg) of paliperidone once daily orally for 24 weeks. Dose adjustment will be done as per Investigator's discretion based upon participant's clinical response to and tolerability of the study drug. Assessments of efficacy will be performed at screening and after 2, 4, 12 and 24 weeks. Efficacy will primarily be evaluated by means of Positive and Negative Syndrome Scale (PANSS). Participants' safety will also be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant meets the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for schizophrenia
* Participant has been given an adequate dose of an appropriate oral atypical antipsychotic for an adequate period of time prior to enrollment, but previous treatment is considered unsuccessful due to one or more of the following reasons: lack of efficacy, lack of tolerability or safety, lack of compliance and/or other reasons to switch to another antipsychotic medication
* Participant or their legally acceptable representatives must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study
* Female participants must be postmenopausal for at least 1 year, surgically sterile, abstinent, or, if sexually active, agree to practice an effective method of birth control before entry and throughout the study and must also have a negative urine pregnancy test at screening
* Male or female, aged greater than or equal to 18 years

Exclusion Criteria:

* Participants on clozapine, any conventional depot neuroleptic or Risperdal CONSTA during the last 3 months
* Participants with serious unstable medical condition, including known clinically relevant laboratory abnormalities
* Participants with history or current symptoms of tardive dyskinesia (twitching or jerking movements that you cannot control in your face, tongue, or other parts of your body)
* Participants with history of neuroleptic malignant syndrome (high fever, rigid muscles, shaking, confusion, sweating more than usual, increased heart rate or blood pressure, or muscle pain or weakness)
* Participants with a current use or known history (over the past 6 months) of substance dependence except for nicotine, caffeine, and betal nut according to DSM-IV Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2008-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan, Ltd. Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone Extended Release (ER): Participants received flexible dose of 3 to 12 milligram (mg) of paliperidone ER once daily orally for 24 weeks. Dose adjustment was done as per Investigator's discretion based upon participant's clinical response to and tolerability of the study drug.
Period: Overall Study
Arm/Group | Paliperidone Extended Release (ER)
Started | 299
Completed | 178
Not Completed | 121
Not completed — Adverse Event | 19
Not completed — Lost to Follow-up | 16
Not completed — Withdrawal by Subject | 25
Not completed — Insufficient Response | 26
Not completed — Ineligible to continue | 8
Not completed — Non-compliant | 9
Not completed — Other | 18

BASELINE CHARACTERISTICS:
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 299
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162
  Male | 137

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 24
Description: The PANSS is a 30-item scale to assess the neuropsychiatric symptoms of schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self). The PANSS provides a total score and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items), each item scored on a scale of 1 (absent) to 7 (extreme). The total score ranges from 30 to 210 and higher score indicates greater severity.
Time Frame: Baseline, Week 24
Population: Intent-to-treat (ITT) population included all participants who received at least 1 dose of study drug and had at least one post-baseline assessment. Missing data was imputed using last observation carried forward (LOCF). Here, 'n' signifies those participants who were evaluable for this outcome measure at specified time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 297
Units on a scale
  Baseline (n=297) | 72.4 (21.1)
  Change at Week 24 (n=281) | -6.9 (17.3)

2. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Marder Subscale Scores at Week 24
Description: The PANSS is a 30-item scale to assess the neuropsychiatric symptoms of schizophrenia. The symptoms are rated on a 7-point scale from 1 (absent) to 7 (extreme psychopathology). Marder PANSS subscales include positive symptoms subscale consisting of 8 items with total score range of 8-56; negative symptoms subscale and disorganized thoughts subscale, each consisting of 7 items with total score range of 7-49; and uncontrolled hostility/excitement (UH/E) subscale and anxiety/depression subscale, each consisting of 4 items with total score range of 4-28. Higher score indicates greater severity.
Time Frame: Baseline, Week 24
Population: ITT population included all participants who received at least 1 dose of study drug and had at least one post-baseline assessment. Missing data was imputed using LOCF. Here, 'n' signifies those participants who were evaluable for this outcome measure at specified time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 297
Units on a scale
  Positive symptoms: Baseline (n=297) | 21.6 (7.2)
  Positive symptoms:Change at Week 24 (n=281) | -2.2 (5.6)
  Negative symptoms: Baseline (n=297) | 17.0 (7.0)
  Negative symptoms:Change at Week 24 (n=281) | -1.7 (4.4)
  Disorganized thoughts: Baseline (n=297) | 16.7 (6.6)
  Disorganized thoughts: Change at Week 24 (n=281) | -1.4 (4.4)
  UH/E: Baseline (n=297) | 7.5 (3.3)
  UH/E: Change at Week 24 (n=281) | -0.5 (3.9)
  Anxiety/depression: Baseline (n=297) | 9.7 (3.8)
  Anxiety/depression:Change at Week 24(n=281) | -1.1 (3.5)

3. Secondary Outcome: Percentage of Participants With at Least 20 Percent Improvement in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: as for outcome 1
Time Frame: Up to Week 24
Population: ITT population included all participants who received at least 1 dose of study drug and had at least one post-baseline assessment. Here 'N' (Number of Participants Analyzed) signifies participants evaluable for this measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 281
Percentage of participants | 31.3

4. Secondary Outcome: Change From Baseline in Total Personal and Social Performance (PSP) Score at Week 24
Description: The PSP is 100-point validated clinician-rated scale that assesses degree of difficulty in 4 areas of functioning: socially useful activities, personal and social relationships, self-care, disturbing and aggressive behaviors rated on 6-point scale (1=absent to 6=very severe).Total transformed score from 1 to 100 is generated from raw score based on clinical interpretation of scores generated in 4 areas of functioning, with higher transformed score indicating better function. Total score is divided into 3 levels: 71-100 (mild difficulty); 31-70 (marked difficulty) and 1-30 (severe difficulty).
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 297
Units on a scale
  Baseline (n=297) | 54.5 (13.8)
  Change at Week 24 (n=269) | 3.4 (12.7)

5. Secondary Outcome: Change From Baseline in Global Assessment of Functioning (GAF) Score at Week 24
Description: The GAF is a 100-point tool rating overall psychological, social and occupational functioning of adults. The higher score range (91-100) refers to a superior functioning in a wide range of activities, and absence of symptoms. The lower score range (1-10) refers to persistent danger of severely hurting self or others; or persistent inability to maintain minimum personal hygiene; or serious suicidal act with clear expectation of death.
Time Frame: Baseline, Week 24
Population: ITT population: all participants who received at least 1 dose of study drug and had at least one post-baseline assessment. Missing data was imputed using LOCF. Here 'N' (Number of Participants Analyzed) signifies number of participants who were evaluable for this measure. 'n' signifies those participants who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 273
Units on a scale
  Baseline (n=273) | 48.9 (14.7)
  Change at Week 24 (n=246) | 5.8 (15.2)

6. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score at Week 24
Description: The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants".
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 297
Units on a scale
  Baseline (n=297) | 4.3 (1.1)
  Change at Week 24 (n=279) | -0.5 (1.1)

7. Secondary Outcome: Change From Baseline in Short-Form 36 Health Survey (SF-36) Score at Week 24
Description: The SF-36 is a health status survey with 36 questions measuring 8 dimensions (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health) that are subsequently aggregated into 2 summary scales, Physical Component Summary (PCS) and Mental Component Summary (MCS). Each item is scored into on a 0-100 range so that the lowest and highest possible scores are set at 0 and 100, respectively. All items are scored so that a high score defines a more favorable health state.
Time Frame: Baseline, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 295
Units on a scale
  PCS: Baseline (n=293) | 61.3 (19.8)
  PCS: Change at Week 24 (n=225) | 0.6 (16.1)
  MCS: Baseline (n=295) | 53.1 (21.5)
  MCS: Change at Week 24 (n=228) | 2.0 (18.4)

8. Secondary Outcome: Number of Participants With Satisfaction With the Study Treatment
Description: Participants assessed their satisfaction with paliperidone ER on a 5-point scale (very good, good, moderate, poor or very poor).
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 237
Participants
  Very good | 11
  Good | 83
  Moderate | 83
  Poor | 49
  Very poor | 11

9. Secondary Outcome: Change From Baseline in Sleep Quality and Daytime Drowsiness Score at Week 24
Description: The Sleep Quality and Daytime Drowsiness evaluation scale is a self-administered scale that rates quality of sleep and daytime drowsiness. Participants indicated on a 5 point scale how well they have slept in the previous 7 days, score ranging from 1 (very badly) to 5 (very well) and how often they have felt drowsy within the previous 7 days, score ranging from 1 (not at all) to 5 (all the time).
Time Frame: Baseline, Week 24
Population: ITT population included all participants who received at least 1 dose of study drug and had at least one post-baseline assessment. Here, 'n' signifies those participants who were evaluable for this outcome measure at specified time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 297
Units on a scale
  Quality of sleep: Baseline (n=297) | 3.2 (1.0)
  Quality of sleep:Change at Week 24 (n=278) | 0.1 (1.1)
  Daytime drowsiness: Baseline (n=297) | 2.6 (1.0)
  Daytime drowsiness:Change at Week 24 (n=278) | -0.3 (1.2)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 24
Arm/Group | Paliperidone Extended Release (ER)
Serious Adverse Events (participants affected / at risk) | 11/299
Other Adverse Events (participants affected / at risk) | 180/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Extended Release (ER) (N=299)
Cellulitis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Blood Electrolytes Abnormal (Investigations) | 1
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemorrhage Intracranial (Nervous system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Delirium (Psychiatric disorders) | 1
Hallucination, Auditory (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Psychotic Disorder (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Extended Release (ER) (N=299)
Palpitations (Cardiac disorders) | 6
Constipation (Gastrointestinal disorders) | 29
Hypersensitivity (Immune system disorders) | 6
Cellulitis (Infections and infestations) | 6
Upper Respiratory Tract Infection (Infections and infestations) | 30
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 11
Akathisia (Nervous system disorders) | 18
Bradykinesia (Nervous system disorders) | 6
Dizziness (Nervous system disorders) | 10
Extrapyramidal Disorder (Nervous system disorders) | 41
Headache (Nervous system disorders) | 14
Parkinsonism (Nervous system disorders) | 8
Sedation (Nervous system disorders) | 10
Somnolence (Nervous system disorders) | 6
Tremor (Nervous system disorders) | 15
Agitation (Psychiatric disorders) | 7
Anxiety (Psychiatric disorders) | 35
Depression (Psychiatric disorders) | 27
Hallucination, Auditory (Psychiatric disorders) | 10
Insomnia (Psychiatric disorders) | 62
Panic Disorder (Psychiatric disorders) | 7
Sleep Disorder (Psychiatric disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dermatitis (Skin and subcutaneous tissue disorders) | 8
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 8

LIMITATIONS AND CAVEATS:
Some Adverse Events summaries were reported based on estimates due to the fact that they were not prepared in the original study report and the relevant definitions of the data elements were not available for these summaries to be regenerated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less